CLINICAL TRIAL: NCT06415760
Title: Reference Range Study for the Quantra System With the QStat Cartridge in Obstetric Patients
Status: Completed | Type: Observational
Sponsor: HemoSonics LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: HEMCS-047
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2025-07-23 (Actual); Status verified 2025-07

CONDITIONS: Obstetric Hemostasis; Coagulation
Keywords: Quantra; Viscoelastic testing; Coagulation
MeSH Terms: conditions — Thrombosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Obstetric Patients: Adult pregnant women in their third trimester of prenancy with no prenatal risk factors and an uncomplicated pregnancy.
  Interventions: Diagnostic Test: Quantra System

INTERVENTIONS:
Diagnostic Test: Quantra System — Diagnostic device to monitor coagulation properties of a whole blood sample at the point-of-care
  Other Names: QStat Cartridge

SUMMARY:
This study will determine reference range intervals for the parameters reported by the Quantra System with the QStat Cartridge in the last trimester of non-laboring pregnant women with an uncomplicated pregnancy

DETAILED DESCRIPTION:
During pregnancy, there is a progressive shift of hemostasis toward a hypercoagulable state that is protective against postpartum hemorrhage. To assess the clinical utility of the Quantra System in high-risk OB patients during delivery, it is important to understand how the normal physiological changes of pregnancy impact Quantra results. This study will determine reference range intervals for the parameters reported by the Quantra System with the QStat Cartridge in the last trimester of non-laboring pregnant women with an uncomplicated pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Subject is female, age 18 to 45 years old.
* Subject is pregnant with a single fetus and duration of pregnancy is >28weeks
* Subject is willing to participate and has provided informed consent.

Exclusion Criteria:

* Subject has a history of a coagulation disorder (including excessive bleeding, thrombosis, VWD, or any factor deficiencies).
* Subject has taken medications known to alter coagulation during pregnancy including heparin, warfarin/Coumadin®, antiplatelet drugs including Plavix® or aspirin at a dose greater than 81 mg/day, Xarelto® or Eliquis®, or other anticoagulants.
* Subject has experienced one or more complications during pregnancy such as gestational diabetes, high blood pressure, pre-eclampsia or eclampsia, hypovolemia or pre-term labor.
* Subject had a blood transfusion during pregnancy.
* Subject has a history of smoking/vaping during pregnancy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: Adult pregnant women 18 years of age or older in their third trimester of pregnancy with no prenatal risk factors and an uncomplicated pregnancy.
Sampling Method: Non-Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2024-05-07 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Reference range intervals for measurement of Clot Stability to Lysis (CSL) parameter | Baseline, determined from a single blood draw
  Reference range intervals for CSL for pregnant women in third trimester
Reference range intervals for measurement of Fibrinogen Contribution (FCS) parameter | Baseline, determined from a single blood draw
  Reference range intervals for FCS for pregnant women in third trimester
Reference range intervals for measurement of Platelet Contribution (PCS) parameter | Baseline, determined from a single blood draw
  Reference range intervals for PCS for pregnant women in third trimester
Reference range intervals for measurement of Clot Stiffness (CS) parameter | Baseline, determined from a single blood draw
  Reference range intervals for CS for pregnant women in third trimester
Reference range intervals for measurement of Clot Time (CT) parameter | Baseline, determined from a single blood draw
  Reference range intervals for CT for pregnant women in third trimester

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - University of Florida Medicine, Gainesville, Florida
  - Unified Womens Clinical Research, Raleigh, North Carolina
  - Unified Womens Clinical Research, Winston-Salem, North Carolina

IPD SHARING:
Plan to Share IPD: No